CLINICAL TRIAL: NCT05870774
Title: Soft Tissue Augmentation Around Implants With Collagen Matrix and Autogenous Graft: 6-months Prospective Randomized Controlled Clinical Trial
Brief Title: Comparative Analysis Using the Collagen Matrix and Autogenous Graft: Clinical Course, Aesthetic Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-02
Record Dates: First submitted 2023-04-25; First posted 2023-05-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2023-04

CONDITIONS: Soft Tissue Atrophy
Keywords: Connective tissue graft; xenogeic collagen matrix; increasing of soft tissue thickness; dental implant; soft tissue augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Active Comparator): The patients underwent implant placement in combination with an increase in the thickness of soft tissues using a free connective tissue graft from the tuberosity area of the upper jaw
  Interventions: Procedure: Soft tissue augmentation with CTG
- Second group (Experimental): The patients underwent implant placement in combination with an increase in the thickness of soft tissues using collagen matrix "Fibro-Gide"
  Interventions: Procedure: Soft tissue augmentation with CM

INTERVENTIONS:
Procedure: Soft tissue augmentation with CTG — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Astra Tech dental implant (Dentsply, Germany)
  3. Harvesting of free connective tissue graft from the maxilla tuberosity area
  4. Fixation of the graft to the vestibular mucosal-periosteal flap
  5. Suturing the wound tightly
  Arms: First group
Procedure: Soft tissue augmentation with CM — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Astra Tech dental implant (Dentsply, Germany)
  3. Modeling of sterile collagen matrix according to the shape of the recipient bed
  4. Fixation of the collagen matrix to the vestibular mucosal-periosteal flap
  5. Suturing the wound tightly
  Arms: Second group

SUMMARY:
This was an interventional prospective randomized clinical trial (RCT) in parallel groups. The sample size is 32 patients who were randomly divided into two groups depending on the surgical intervention used. First group - patients underwent increasing the thickness of the mucous membrane using free connective tissue graft from tuberosity area of the upper jaw. Second group - patients used collagen matrix Fibro-Gide" (Geistlich Pharma AG, Bahnhofstrasse 40, 6110 Wolhusen, Switzerland; registration in Russia 19.08.2020 No FSZ -20207/11765). In the postoperative period the value of soft tissue thickness gain, severity of pain, collateral edema, amount of analgesics consumed, soft tissue aesthetics, keratinized mucosa width, quality of life and duration of surgery were assessed.

DETAILED DESCRIPTION:
The aim of this research was to perform a comparative clinical analysis of soft tissues in the area of soft tissue graft and collagen matrix transplantation. Thirty two patients diagnosed with partial absence of teeth was examined on the basis of the Department of Surgical Dentistry of the E.V. Borovsky Institute of Dentistry of I.M. Sechenov First Moscow State Medical University. Patients had a soft tissue thickness deficiency from the vestibular surface in the area of the planned dental implant placement in the distal parts of the mandible, which was an indication for its increase. All patients were randomly divided into two groups depending on method of soft tissue augmentation used. In 1 group (n=16) transplantation of a free connective tissue graft (CTG) from tuberosity area of the upper jaw was performed. In 2 group (n=16) collagen matrix "Fibro-Gide" was used. According to gender and age characteristics, both groups were comparable. Randomization of patients was carried out at the stage of surgical intervention as follows: after a dental implant placement and preparation of recipient's bed, an envelope with a randomly assigned treatment method (using a connective tissue graft or a collagen matrix) was opened.

During the operation, incision was made along the top of the alveolar ridge within the defect; a full-thickness muco-periosteal flap was elevated. Traditional 2-stage dental implantation was performed according to surgical protocols of dental implant systems Astra Tech (Dentsply Implants Manufacturing GmbH, Germany; registration in Russia 27.12.2019 No FSZ 2015/3214). A free connective tissue graft was harvested in patients of the first group. Graft was fixed with a horizontal U-shaped suture to the buccal muco-periosteal flap. In second patients group a fragment of the collagen matrix "Fibro-Gide" was fixed to the buccal muco-periosteal flap (Geistlich Pharma AG, Bahnhofstrasse 40, 6110 Wolhusen, Switzerland; registration in Russia 19.08.2020 No FSZ - 20207/11765). For patients of all groups mobilization of the muco-periosteal flap conducted followed by suturing the wound tightly without tension with simple interrupted sutures.

Postoperative recommendations included standard antibacterial and anti-inflammatory therapy in combination with the use of local antiseptics for daily care was prescribed.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of written informed consent of the patient to participate in the study;
2. Age from 25 to 59 years;
3. The presence of an included defect in the distal part of the lower jaw with a sufficient volume of bone tissue;
4. Soft tissue thickness <3 mm on the vestibular side;
5. Adjacent teeth without periodontal pathology, the depth of probing should not exceed 3 mm along the entire dentoalveolar furrow;
6. Satisfactory level of oral hygiene;
7. Patients without concomitant pathology or with concomitant pathology in the compensation stage.

Non-inclusion criteria:

1. Age less than 25 and more than 59 years;
2. Hard smokers (more than 10 cigarettes a day);
3. The presence of concomitant pathology in the stage of decompensation;
4. Patients with malignant tumors, as well as patients with a history of radiation and chemotherapy over the past 5 years;
5. Taking medications that affect the healing of soft tissues (nonsteroidal anti-inflammatory drugs, steroid drugs);
6. Pregnancy and breastfeeding;
7. Patients with mental disorders.

Exclusion Criteria:

1. Patients with infections either periodontally or periapically, which developed after inclusion in the study;
2. Pregnancy following entrance into the study;
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures;
4. Patients who, for one reason or another, could not complete the entire protocol to the end.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
The amount of soft tissue thickness gain | [Day 90 compared to the 0th day (initial value)]
  The value of soft tissue thickness gain in the study area (mm) on the 90th day compared to the 0th day (initial value).To carry out the measurement an optical impression was taken using the Primescan intraoral scanner (Dentsply/SIRONA,Germany, 16.05.2019, № RD-27221/26851) before the operation and on the 90th day after the operation. Further, in the specialized program GOM Inspect the stl-files were compared and the vestibular contour changes were evaluated at 3 equidistant points in the coronary-apical direction. The мean value between the points was the amount of soft tissue thickness gain (mm).

SECONDARY OUTCOMES:
The amount of soft tissue thickness gain | [Day 180 compared to the 0th day (initial value)]
  The value of soft tissue thickness gain in the study area (mm) on the 180th day compared to the 0th day (initial value).To carry out the measurement an optical impression was taken using the Primescan intraoral scanner (Dentsply/SIRONA,Germany, 16.05.2019, № RD-27221/26851) before the operation and on the 180th day after the operation. Further, in the specialized program GOM Inspect the stl-files were compared and the vestibular contour changes were evaluated at 3 equidistant points in the coronary-apical direction. The мean value between the points was the amount of soft tissue thickness gain (mm).
Assessment of the severity of pain syndrome | [Day 1 compared to the 0th day (initial value)].
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [Day 3 compared to the 0th day (initial value)].
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [Day 5 compared to the 0th day (initial value)].
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [Day 7 compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [Day 90 compared to the 0th day (initial value)].
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [Day 180 compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the collateral edema | [Day 1 compared to the 0th day (initial value)].
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | [Day 3 compared to the 0th day (initial value)].
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | [Day 5 compared to the 0th day (initial value).]
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | [Day 7 compared to the 0th day (initial value).]
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of consumption of analgesics | [Day 1 compared to the 0th day (initial value).]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of consumption of analgesics | [Day 3 compared to the 0th day (initial value).]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of consumption of analgesics | [Day 5 compared to the 0th day (initial value).]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of consumption of analgesics | [Day 7 compared to the 0th day (initial value).]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of the quality of life | [Day 7 compared to the 0th day (initial value).]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.
Assessment of the quality of life | [Day 90-93 compared to the 0th day (initial value).]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.
Assessment of the quality of life | [Day 180-186 compared to the 0th day (initial value).]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.
Attached mucosa measurement | [Day 0 (initial value)]
  The width of the keratinised attached mucosa was measured using the UNC-15 periodontal probe. This was done by determining the mucosa-gingival junction line on the vestibular side. The distance from this line to the apex of the alveolar ridge was correspond to the width of the keratinised attached mucosa.
Attached mucosa measurement | [Day 90-93 compared to the 0th day (initial value)].
  The width of the keratinised attached mucosa was measured using the UNC-15 periodontal probe. This was done by determining the mucosa-gingival junction line on the vestibular side. The distance from this line to the apex of the alveolar ridge was correspond to the width of the keratinised attached mucosa.
Attached mucosa measurement | [Day 180-186 compared to the 0th day (initial value)].
  The width of the keratinised attached mucosa was measured using the UNC-15 periodontal probe. This was done by determining the mucosa-gingival junction line on the vestibular side. The distance from this line to the apex of the alveolar ridge was correspond to the width of the keratinised attached mucosa.
Soft tissue aesthetics | [Day 180-186 compared to the 0th day (initial value) ]
  Evaluation of soft tissue aesthetics was carried out by visual inspection taking into account the PES (pink aesthetic score). The evaluation was carried out according to a score of 0-1-2, where 0 was the lowest value and 2 was the highest, the maximum achievable PES value was 14.
Microbiota Evaluation | [Day 90]
  At 3 months, mucosal swabs from the implant emergence profile were collected and transported in Amies medium. Samples were cultured on selective and blood agar under aerobic and anaerobic conditions. Colonies were counted and identified using biochemical tests and MALDI-TOF mass spectrometry (score ≥2.0 considered reliable). Species diversity with clinically significant growth (CFU/mL ≥ 105); microbiome formation duration (p=0.04131); the expression of the TNFα gene were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Ashurko, ass.prof., Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (1):
- I.M. Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashurko I, Tarasenko S, Magdalyanova M, Balyasin M, Galyas A, Kazumyan S, Safi N, Unkovskiy A. 3D-Analysis of Peri-Implant Soft Tissue Gain With Collagen Matrix and Connective Tissue Graft: A Randomized Control Trial. Clin Implant Dent Relat Res. 2025 Apr;27(2):e70043. doi: 10.1111/cid.70043. PMID 40254798